CLINICAL TRIAL: NCT01503684
Title: Biomarkers in Exhaled Breath Condensates of Septic Patients to Predict Development of Multi-organ Dysfunction Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201106068RC
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2011-09

CONDITIONS: Sepsis
Keywords: sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath condensate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with sepsis: Patients who are admitted to ICU with the diagnosis of sepsis
  Interventions: Other: Determined by intended physician

INTERVENTIONS:
Other: Determined by intended physician — We perform a prospective observational study. All the treatment for the patients are determined by intended physicians.

SUMMARY:
In this proposal, the investigators wish to investigate, identify and validate potential biomarkers in collected exhaled breath condensates (EBC) from patients with sepsis.

DETAILED DESCRIPTION:
In this proposed project, we will focus on the identification of potential biomarkers in EBC with ability to predict development of multi-organ failure. Currently, no tools could be used to evaluate the effect of mitochondrial dysfunction in sepsis. All the human studies discussing mitochondrial dysfunction in sepsis use tissue biopsies as study materials. Repeated tissue biopsy is invasive and not applicable. EBC could be collected non-invasively and conveniently. A study has demonstrated the use of metabolomic technologies in mitochondrial diseases. We believe that the metabolomic biomarkers of EBC could be used to demonstrate mitochondrial dysfunction in lungs and respiratory tracts of septic patients. Such metabolomic biomarkers may also reflect similar on-going mitochondrial dysfunction in other organ systems, and could potentially become a novel diagnostic tool and a therapeutic target in future sepsis therapy.

ELIGIBILITY:
Inclusion Criteria:

* above 20 years old
* admitted to ICU with the diagnosis of sepsis and treated with mechanical ventilation via an endotracheal tube

Exclusion Criteria:

* pregnant
* active malignancy
* in an immunosuppressed status such as HIV disease, neutropenia, being treated with immunosuppressive agents
* expected to have an unavoidable very short life expectancy after admission, i.e., < 3 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to ICU with the diagnosis of sepsis and treated with mechanical ventilation via an endotracheal tube.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-08

PRIMARY OUTCOMES:
Development and severity of sepsis | 28 days
  To record APACHE II, SOFA, and MODS, etc.

SECONDARY OUTCOMES:
Mortality | 28 days
Response to treatment and progression of organ failure | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Shuin Jerng, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan